CLINICAL TRIAL: NCT07328659
Title: Our Stone Fixation Technique to Improve the Efficacy of Peumatic Lithotripsy With Suction Sheath in Mini-pcnl.
Brief Title: Our Study About Anew Technique to Improve Results of Peumatic Lithotripsy in Mimi Pcnl With Suction Sheath.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yasser Gamil Elnagar (Other)
Responsible Party: Sponsor-Investigator, Yasser Gamil Elnagar, Principal Investigator, Aswan University
Organization: Aswan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAD-MC-2025-001
Record Dates: First submitted 2025-12-06; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Kidney Stone; Calculi, Renal
Keywords: Urolithiasis; Endourology; Suction sheath
MeSH Terms: conditions — Kidney Calculi; Urolithiasis

STUDY DESIGN:
Intervention Model Description: Single group quasi interventional prospective study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with kidney stones treated by our technique (Experimental): Prospective assesment of results.
  Interventions: Procedure: Peumatic lithotripsy in mini-pcnl

INTERVENTIONS:
Procedure: Peumatic lithotripsy in mini-pcnl — Using our technique to improve results of peumatic lithotripsy in suction mini-PCNL.

SUMMARY:
Prospective study to assist safty and efficieny of our technique of using peumatic lithotripsy with suction mini-pcnl.

DETAILED DESCRIPTION:
anew techniqe was designed to improve the results of pneumatic lithotripsy in suction mini-PCNL by:

1. Customize our instrument to be suitable for a short 12 Fr nephroscope.
2. using certain measures to avoid stone migration during pneumatic disintegration.

By fixing stones during disintegration and suction.

* Our puncture strategy was planned to prevent stone migration.
* Use a suction sheath to gently fix the stone between the tip of the sheath and the inner wall of the kidney and disintegrate it from inside the sheath.
* The dormai basket was used to fix the stone in front of the sheath in difficult situations.

The investigators will assess disintegration time as the primary endpoint and stone-free rate and complications as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* any patient with kidney stones less than 4 cm .

Exclusion Criteria:

* children less than 3 yrs.
* single kidney patient.
* patient with ectopic kidney and spinal deformities.
* unfit patient for surgry.

Ages: 3 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Stone disintegration time | Day 1
  Assesment of peumatic lithotripsy time during the operation.

SECONDARY OUTCOMES:
Stone free rate | -after the operation immediately and then after 1 month of the operation.
  Presence of residual stones more than 3mm
Rate of complications | Intraoperative and immediately post operative till one week.
  rate of any intra or postoperative coplications.

CONTACTS AND LOCATIONS:
Locations (1):
- Radar medical centre, Aswān, Aswan Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No